CLINICAL TRIAL: NCT06379061
Title: Access MeMed BV Assay Clinical Study Collection Protocol - Infectious Adult and Pediatric Cohorts
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MM-01-24; MMP-01-24 (Other: Beckman Coulter, Inc.)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Infection, Bacterial; Infection Viral
MeSH Terms: conditions — Bacterial Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma Specimens fully de-identified
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult and Pediatrics: A minimum of 244 serum samples will be collected at a minimum of two (2) US locations from enrolled pediatric and adult patients presenting signs and symptoms suggestive of acute bacterial or viral infection. The number of patients enrolled is based on total volume required to run analytical comparison studies under a future testing protocol.
  Interventions: Other: Adult and Pediatrics

INTERVENTIONS:
Other: Adult and Pediatrics — This is an observational study. This protocol is for blood draw enrollment. These samples will be collected and binned by their results from the MeMed BV assay. Samples collected will be used for an analytical comparison study under a future testing protocol. These samples will be used to establish the diagnostic performance of MeMed BV test on BEC Access Immunoassay Systems for differentiating bacterial from viral infection.

SUMMARY:
The purpose of the pivotal study is to collect blood specimens and clinical data from pediatric (>90 days old) and adult (≥18 years old) patients presenting with signs and symptoms suggestive of acute bacterial or viral infection. These samples will be used to establish the diagnostic performance of MeMed BV™ for differentiating bacterial from viral infection using method comparison and/or method concordance.

DETAILED DESCRIPTION:
The objective of this study is to collect blood specimens from pediatric (>90 days old) and adult patients (≥18 years old) presenting with signs and symptoms suggestive of acute bacterial or viral infection from hospital, Emergency Department, or Urgent Care Centers for comparative testing on the Access 2 and DxI 9000 Immunoassay Analyzers.

ELIGIBILITY:
Inclusion Criteria:

* Over 90 days of age.
* Clinical suspicion of acute bacterial or viral infection.
* Temperature ≥ 37.8°C (100°F) (any body site, any measurement device, including self-reported) or tactile fever, either of them noted at least once within the last 7 days.
* Current disease duration ≤ 7 days.

Exclusion Criteria:

* Previously enrolled
* Insufficient sample volumes obtained

  * For the adult and pediatric populations, < 1.2 mL serum volume
* Sample handling errors
* Another unrelated episode of febrile infection within the past 2 weeks
* Suspicion and/or confirmed diagnosis of infectious gastroenteritis/ colitis.
* ≥48 hours of oral antibiotic treatment
* ≥12 hours of intravenous\intramuscular antibiotic treatment
* Human Immunodeficiency Viruses (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (self-declared or known from medical records)
* A proven or suspected infection on presentation with Mycobacterial (e.g., Tuberculosis, MAC), parasitic or fungal (e.g., Candida, Histoplasma, Aspergillus) pathogen
* Active inflammatory disease (e.g., Inflammatory Bowel Disease [IBD], Systemic Lupus Erythematosus [SLE], Juvenile Idiopathic Arthritis [JIA], Rheumatoid Arthritis [RA], Kawasaki, other vasculitis)
* Major trauma and\or burns in the last 7 days.
* Major surgery in the last 7 days
* Congenital immune deficiency (CID)
* Acquired immune deficiency\modulation state including

  1. Active malignancy treated within last 6 months
  2. Current treatment with immune-suppressive or immune-modulating therapies, including without limitations:

  i. Administration of P.O.\IV\IM high dose steroids >1mg/kg/day prednisone (or equivalent) at some point in the past 10 days or daily continuous use of steroids > 0.25 mg/kg/day in the past 7 days ii. Monoclonal antibodies, anti-TNF agents iii. Intravenous immunoglobulin (IVIG) iv. Cyclosporine, Cyclophosphamide, Tacrolimus, Azathioprine, Methotrexate v. G/GM-CSF Interferons c. Post solid organ/bone marrow transplant patients d. Asplenia, sickle cell disease
* Indwelling central venous catheter
* Cystic Fibrosis
* Pregnancy - self-reported or medically known
* Other severe illnesses that affect life expectancy and quality of life such as:

  1. Severe psychomotor retardation
  2. Congenital metabolic disorder
  3. End stage renal disease, advanced heart failure (NYHA 3/4), advanced COPD (GOLD 3/4)

Ages: 90 Days to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients presenting to the Emergency Department or Urgent Care Center with signs and symptoms suggestive of acute bacterial or viral infection.
  The study sample size will be divided into the following:
  * Pediatric (>90 days - <18 yrs. of age) population sample target of 30 enrolled subjects.
  * Adult (≥18 yrs. of age) population sample target of 214 adult patients enrolled subjects.
  The target population will be representative of US demographics. This sample size aligns with comparator device studies. Pediatric sample collection will be separated into the following three (3) age categories:
  * Age over 90 days to <2 yrs.
  * Age 2 yrs. to <12 yrs.
  * Age 12 yrs. to <18 yrs.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Blood Specimen Collection | Less or equal to seven days
  Collect blood specimens across multiple age ranges presenting symptoms of acute or viral infection

CONTACTS AND LOCATIONS:
Overall Officials: David Haan, Study Director — Beckman Coulter, Inc.
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Brigham, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No